CLINICAL TRIAL: NCT04759300
Title: Effectiveness of C-MAC Video-stylet Versus C-MAC D- Blade Video-laryngoscope for Tracheal Intubation in Patients With Predicted Difficult Airway: Randomized Comparative Study
Brief Title: Effectiveness of C-MAC Video-stylet Versus C-MAC D- Blade Video-laryngoscope for Tracheal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, rehab zayed, Assisstant Professor of Anesthesia, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0304844
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Difficult Mask Ventilation; Difficult Intubation

STUDY DESIGN:
Intervention Model Description: The patients will be randomly assigned into two equal groups using computer-generated randomization technique. Group C-MAC VS (VS group) included patients undergoing tracheal intubation using the C-MAC VS. Group C-MAC VL D -blade (D group) included patients undergoing intubation using the C-MAC VL D-blade.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C-MAC VS (Active Comparator): patients undergoing tracheal intubation using the C-MAC VS.
  Interventions: Device: C-MAC VS
- Group C-MAC VL D -blade (Placebo Comparator): patients undergoing intubation using the C-MAC VL D-blade.
  Interventions: Device: C-MAC VL D -blade

INTERVENTIONS:
Device: C-MAC VS — patients undergoing tracheal intubation using the C-MAC VS
  Arms: Group C-MAC VS
Device: C-MAC VL D -blade — patients undergoing intubation using the C-MAC VL D-blade.
  Arms: Group C-MAC VL D -blade

SUMMARY:
Videolaryngoscopy provides a better laryngeal view and do not need airway alignment for tracheal intubation.

DETAILED DESCRIPTION:
The C-MAC-VS can be connected easily to the same C- MAC monitor and Pocket Monitor without requiring any additional light source and camera. This device is great for cases with limited mouth opening, airway obstruction and difficult intubation. C-MAC-VS has no lumens so it's very easy to clean and it can accommodates a size ETT 6.0 and greater.

ELIGIBILITY:
Inclusion Criteria:

* patients with BMI ≥ 30 kg/m2,
* presence of any predictors of difficult intubation;
* Mallampati score > =3;
* inter-incisor distance < 3 cm;
* thyromental distance < 6 cm;
* neck extension < 80°from neck flexion;
* cervical spine instability; history of difficult endotracheal intubation or difficult mask ventilation

Exclusion Criteria:

* patients have increased risk of pulmonary aspiration;
* have significant medical diseases in term of cardiac, respiratory, hepatic, renal

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
duration of intubation procedure | 10 minutes
  assess duration of intubation procedure by using C-MAC VS versus C-MAC D-blade in patients with anticipated difficult airway.

CONTACTS AND LOCATIONS:
Overall Officials: rehab A. Abd Elaziz, Ass.Prof., Principal Investigator — Alexandria University
Locations (1):
- rehab Abd Elaziz, Alexandria, Egypt